CLINICAL TRIAL: NCT01672307
Title: Efficacy and Tolerability of Minoxidil 2% for Eyebrow Enhancement : A Randomized , Double-blind , Placebo-controlled , Split-face Comparative Study
Brief Title: Minoxidil 2% for Eyebrow Enhancement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mae Fah Luang University Hospital (Other)
Responsible Party: Principal Investigator, Chuchai TANGLERTSAMPAN, MD, Instructor, Mae Fah Luang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MFL University
Record Dates: First submitted 2012-08-19; First posted 2012-08-24 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Hypotrichosis of Eyebrows; Thinning Eyebrows
Keywords: hypotrichosis of eyebrows; thinning eyebrows; minoxidil; placebo; randomized

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minoxidil lotion 2% (Experimental): Minoxidil lotion 2% is applied twice daily to one eyebrow.
  Interventions: Drug: Minoxidil lotion 2%
- Placebo (Placebo Comparator): Placebo is applied twice daily to the other eyebrow.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minoxidil lotion 2% — Minoxidil lotion 2% is applied twice daily to one eyebrow.
  Arms: Minoxidil lotion 2%
Drug: Placebo — Placebo is applied twice daily to the other eyebrow.
  Arms: Placebo

SUMMARY:
The purpose of the study is to compare minoxidil 2% versus placebo in enhancement of eyebrows.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged 18-40 years
* hypotrichosis of eyebrows
* healthy
* informed consent obtained

Exclusion Criteria:

* no underlying diseases
* no alopecia areata or trichotillomania
* no thyroid diseases
* no pregnancy or breast feeding
* no previous eyebrow tattoo, trauma or accident.
* no history of eyebrow or hair medications in 6 months
* no history of minoxidil or its ingredient allergy
* no history of eyebrow surgery.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The change of global photographic assessment after 16 weeks from baseline | baseline and 16 weeks

SECONDARY OUTCOMES:
The change of hair diameter after 16 weeks from baseline | baseline and 16 weeks

OTHER OUTCOMES:
The change in number of hairs after 16 weeks from baseline | baseline and 16 weeks
Number of participants with adverse events. Adverse events include any skin rashes or symptoms. | 16 weeks
Patient satisfaction by self-assessment questionnaires | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chuchai Tanglertsampan, MD, Principal Investigator — MFL University Hospital (Bangkok)
Locations (1):
- MFL University Hospital (Bangkok), Bangkok, Thailand